CLINICAL TRIAL: NCT06847464
Title: A Non-Randomized, Open-Label, Drug-Drug Interaction Study to Evaluate the Effects of Itraconazole, Carbamazepine, Quinidine, and Fluconazole on the Pharmacokinetics and Safety of EDP-323 in Healthy Participants
Brief Title: A Drug-Drug Interaction Study to Evaluate the Effects of Itraconazole, Carbamazepine, Quinidine and Fluconazole on the Pharmacokinetics and Safety of EDP-323.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 323-005
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: RSV Infection; Drug Drug Interaction (DDI)
Keywords: Drug Drug Interaction
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Itraconazole; Carbamazepine; Quinidine; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- EDP-323 and itraconazole interaction (Part 1) (Experimental): Subjects will receive EDP-323 and itraconazole on respective dosing days
  Interventions: Drug: EDP-323; Drug: Itraconazole
- EDP-323 and carbamazepine interaction (Part 2) (Experimental): Subjects will receive EDP-323 and carbamazepine on respective dosing days
  Interventions: Drug: EDP-323; Drug: carbamazepine
- EDP-323 and quinidine interaction (Part 3) (Experimental): Subjects will receive EDP-323 and quinidine on respective dosing days
  Interventions: Drug: EDP-323; Drug: Quinidine
- EDP-323 and fluconazole interaction (Part 4) (Experimental): Subjects will receive EDP-323 and fluconazole on respective dosing days
  Interventions: Drug: EDP-323; Drug: fluconazole

INTERVENTIONS:
Drug: EDP-323 — Subjects will receive EDP-323 on Days 1 and 14
  Arms: EDP-323 and itraconazole interaction (Part 1)
Drug: Itraconazole — Subjects will receive itraconazole QD Days 5-18
  Arms: EDP-323 and itraconazole interaction (Part 1)
Drug: EDP-323 — Subjects will receive EDP-323 on Days 1 and 23
  Arms: EDP-323 and carbamazepine interaction (Part 2)
Drug: carbamazepine — Subjects will receive carbamazepine on Days 5 - 27
  Arms: EDP-323 and carbamazepine interaction (Part 2)
Drug: EDP-323 — Subjects will receive EDP-323 on Days 1 and 8
  Arms: EDP-323 and quinidine interaction (Part 3)
Drug: Quinidine — Subjects will receive quinidine on Days 5-12
  Arms: EDP-323 and quinidine interaction (Part 3)
Drug: EDP-323 — Subjects will receive EDP-323 on Days 1 and 14
  Arms: EDP-323 and fluconazole interaction (Part 4)
Drug: fluconazole — Subjects will receive fluconazole on Days 5-18
  Arms: EDP-323 and fluconazole interaction (Part 4)

SUMMARY:
The primary aim of the study is to assess the effect of itraconazole, carbamazepine, quinidine, and fluconazole individually on the pharmacokinetics and safety of EDP-323 in healthy adult participants. Each participant's duration in the study will be dependent upon which study part they are enrolled.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 65 years, inclusive.
* Screening body mass index (BMI) of 18 to 30 kg/m2 with a minimum body weight of50 kg
* Female subjects of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 30 days after the last dose of EDP-323. A male participant who has not had a vasectomy and is sexually active with a woman of childbearing potential must agree to use effective contraception from the date of Screening to 90 days after his last dose of study drug.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease
* Pregnant or nursing females
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection
* A positive urine drug screen at Screening or Day -1
* Current tobacco smokers or use of tobacco within 3 months prior to Screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy)
* History of regular alcohol consumption exceeding protocol limits
* Participation in a clinical trial within 28 days prior to the first dose of study drug
* For Part 2 and Part 3 participants, the following cardiovascular abnormalities:
* QRS duration >110 ms
* Incomplete right bundle branch block or any complete bundle branch block
* Heart rate <40 or >90 beats per minute (per vital sign capture while rested)
* History of unexplained syncope, structural heart disease, or clinically significant arrhythmias
* Personal or family history of long QT syndrome (genetically proven or suggested by sudden death of a close relative due to cardiac causes at a young age) or Brugada syndrome
* PR interval >220 ms or any 2nd or 3rd degree AV block
* Ventricular pre-excitation
* Other exclusions for Part 2 (carbamazepine) participants
* Participants of Asian ancestry with HLA allele B*1502 in this population
* Platelets, white blood cell count or hemoglobin below the lower limit of normal, due to reported incidence of agranulocytosis and aplastic anemia with carbamazepine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-05-24 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP-323 with and without coadministration with Itraconazole | Day 1 through Day 19
AUC of EDP-323 with and without coadministration with Itraconazole | Day 1 through Day 19
Cmax of EDP-323 with and without coadministration with Carbamazepine | Day 1 through Day 28
AUC of EDP-323 with and without coadministration with Carbamazepine | Day 1 through Day 28
Cmax of EDP-323 with and without coadministration with Quinidine | Day 1 through Day 13
AUC of EDP-323 with and without coadministration with Quinidine | Day 1 through Day 13
Cmax of EDP-323 with and without coadministration with fluconazole | Day 1 through Day 19
AUC of EDP-323 with and without coadministration with fluconazole | Day 1 through Day 19

SECONDARY OUTCOMES:
Safety measured by adverse events | Up to 34 Days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- ICON, plc, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No